CLINICAL TRIAL: NCT05587491
Title: Feasibility and Safety of HybridAPC for Gastric Mucosal Ablation in the Management of Patients With Obesity.
Brief Title: HybridAPC for Gastric Mucosal Ablation in Obese Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erbe Elektromedizin GmbH (Industry)
Collaborators: ERBE AUSTRALIA PTY LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021_03
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Adiposity
Keywords: Endoscopic bariatric therapy; Hybrid Argonplasma Coagulation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric mucosal ablation (Other): Participants receive submucosal injection followed by ablation of gastric mucosa using Hybrid argonplasma.
  Interventions: Device: Hybrid Argonplasma coagulation (HAPC)

INTERVENTIONS:
Device: Hybrid Argonplasma coagulation (HAPC) — Gastric mucosal ablation is an endoscopic procedure which uses argonplasma coagulation in combination with submucosal injection to achieve selective ablation

SUMMARY:
This study is intended to investigate safety and feasibility of a new weight loss technique called Gastric Mucosal Ablation (GMA) that does not require surgery, but can be achieved using an endoscopic procedure.

Previous studies have suggested that weight loss after vertical sleeve gastrectomy (VSG) is partly due to the removal of normal stomach tissue suspected of having hormonal function. The study will investigate the minimally invasive treatment of obese participants by means of argon plasma coagulation (APC) in combination with waterjet submucosal injection using HybridAPC.

As primary endpoint the % total body weight loss (TBWL) will be determined as body weight difference at the final 6 months FU after the last treatment session in comparison to the body weight prior to the initial treatment.

After signing the informed consent the doctor and research team will determine if the participant meets all requirements for this study. If a participant is confirmed to be a suitable candidate additional tests will be performed prior to the first application of GMA to assess the health status of the participant prior to treatment. During the screening and baseline visit the medical history and the medications of the participant will be reviewed.

After the treatments the participants will be followed for up to 6 months to assess the outcome of the GMA procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females patients in the range of class I to class III obesity (30 ≤ BMI ≤ 45).
2. Age 21 - 75 yrs.
3. Treatment naïve for bariatric surgery or endoscopic bariatric therapy
4. Agree to avoid any use of weight loss medications such as Meridia, Saxenda, Januvia, Xenical, or over the counter weight loss medications or supplements throughout the study.
5. Women of childbearing potential (WOCBP) must agree to use acceptable contraception methods.
6. Agree not to donate blood during their participation in the study.
7. Able to comply with study requirements and understand and sign the Informed Consent Form.
8. Stable weight defined as a fluctuation of less than 5% for at least 3 months prior to screening visit.

Exclusion Criteria:

1. Patients requiring exogenous insulin.
2. HbA1c > 9.5 %
3. Pregnant or breast-feeding or intending to get pregnant during the study.
4. Unwilling or unable to complete the patient diary, or comply with study visits and other study procedures as required per protocol.
5. History of diabetic ketoacidosis or hyperosmolar nonketotic coma.
6. Probable insulin production failure, defined as fasting C-Peptide serum < 1 ng/mL (333 pmol/l).
7. Previous use of any types of insulin for > 1 month (at any time, except for treatment of gestational diabetes).
8. Change in diabetic treatment within the last three months.
9. Use of glucose-lowering drugs for diabetes mellitus treatment with the exception of sulfonylurea (SU), biguanides and sodium dependent glucose co-transporter 2 (SGLT-2) inhibitors.
10. Change of diabetes medication or doses 12 weeks prior to screening visit.
11. Hypoglycemia unawareness or a history of severe hypoglycemia (more than 1 severe hypoglycemic event, as defined by need for third-party-assistance, in the last year).
12. Known autoimmune disease, including but not limited to celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder.
13. Previous upper GI surgery, or other endoscopic bariatric procedures or conditions, prior intra-gastric balloon or another gastric implant.
14. History of diabetic gastroparesis.
15. Known active hepatitis or active liver disease.
16. Acute gastrointestinal illness in the previous 7 days.
17. Known history irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease.
18. Known history of a structural or functional disorder of the esophagus that may impede passage of the device through the gastrointestinal tract or increase risk of esophageal damage during an endoscopic procedure, including Barrett's esophagus, esophagitis, dysphagia, achalasia, stricture/stenosis, esophageal varices, esophageal diverticula, esophageal perforation, or any other disorder of the esophagus.
19. Known history of a structural or functional disorder of the esophagus, including any swallowing disorder, esophageal chest pain disorders, or drug refractory esophageal reflux symptoms.
20. Known history of a structural or functional disorder of the stomach including gastroparesis, gastric ulcer, chronic gastritis, gastric varices, hiatal hernia (>3 cm), cancer or any other disorder of the stomach.
21. Known history of chronic symptoms suggestive of a structural or functional disorder of the stomach, including any symptoms of chronic upper abdominal pain, chronic nausea, chronic vomiting, chronic dyspepsia or symptoms suggestive of gastroparesis, including post-prandial fullness or pain, post-prandial nausea or vomiting or early satiety.
22. Currently have ongoing symptoms suggestive of intermittent small bowel obstruction, such as recurrent bouts of post-prandial abdominal pain, nausea or vomiting.
23. Active H. pylori infection (Subjects with active H. pylori may continue with the screening process if they are treated with an appropriate antibiotic regimen, and eradication has been confirmed).
24. History of coagulopathy, upper gastrointestinal bleeding conditions such as ulcers, gastric varices, strictures, congenital or acquired intestinal telangiectasia.
25. Current use of anticoagulation therapy
26. Obligate use of anti-inflammatory drugs that cannot be suspended for a minimum of 4 weeks post procedure
27. Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit.
28. Use of drugs known to affect GI motility (e.g. Metoclopramide).
29. Receiving any weight loss medications such as Meridia, Xenical, Saxenda, Januvia, Duromine or over the counter weight loss medications at screening.
30. Untreated/inadequately treated hypothyroidism, defined as an elevated Thyroid-Stimulating Hormone (TSH) level at Screening; if on thyroid hormone replacement therapy, must be on stable dose for at least 6 weeks prior to Screening.
31. Persistent Anemia, defined as Hemoglobin <10 g/dL.
32. Subjects who have donated blood or received a transfusion in the prior 3 months.
33. Subjects with conditions that alter red blood cell turnover.
34. Significant cardiovascular disease including known history of valvular disease, or myocardial infarction, heart failure, transient ischemic attack or stroke within the last 6 months.
35. Moderate or severe chronic kidney disease (CKD), with estimated glomerular filtration rate (eGFR) <45 ml/min/1.73m2 (estimated by MDRD).
36. Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy or radiotherapy within the past 12 months, who have clinically-significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the subject a poor candidate for clinical trial participation in the opinion of the Investigator.
37. Active systemic infection.
38. Active malignancy within the last 5 years (with the exception of treated basal cell or treated squamous cell carcinoma).
39. Subjects with an established diagnosis of Multiple Endocrine Neoplasia syndrome type 1.
40. Not a candidate for surgery or general anesthesia.
41. Active illicit substance abuse or alcoholism.
42. Current smoker or smoking history in the last six months.
43. Participating in another ongoing clinical trial of an investigational drug or device.
44. Any other mental or physical condition which, in the opinion of the Investigator, makes the subject a poor candidate for clinical trial participation.
45. Other medical condition that does not allow for endoscopic procedure.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Assessment of the % of total body weight loss (% TBWL). | 9 months
  TBWL will be determined as body weight difference at the final 6 months FU after the last treatment session in comparison to the body weight prior to the initial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Sartoretto, MBBS, BMedSc, Principal Investigator — The Bariatric & Metabolic Institute The BMI Clinic, Australia
Locations (1):
- The Bariatric & Metabolic Institute The BMI Clinic, Double Bay, New South Wales, Australia

REFERENCES:
- [Background] Oberbach A, Schlichting N, Heinrich M, Kullnick Y, Retschlag U, Lehmann S, Khashab MA, Kalloo AN, Kumbhari V. Gastric mucosal devitalization reduces adiposity and improves lipid and glucose metabolism in obese rats. Gastrointest Endosc. 2018 Jan;87(1):288-299.e6. doi: 10.1016/j.gie.2017.04.038. Epub 2017 May 4. PMID 28479494
- [Background] Kumbhari V, Lehmann S, Schlichting N, Heinrich M, Kullnick Y, Retschlag U, Enderle M, Dietrich A, Khashab MA, Kalloo AN, Oberbach A. Gastric mucosal devitalization is safe and effective in reducing body weight and visceral adiposity in a porcine model. Gastrointest Endosc. 2018 Jul;88(1):175-184.e1. doi: 10.1016/j.gie.2018.02.022. Epub 2018 Feb 22. PMID 29476845
- [Background] Fayad L, Oberbach A, Schweitzer M, Askin F, Voltaggio L, Larman T, Enderle M, Hahn H, Khashab MA, Kalloo AN, Kumbhari V. Gastric mucosal devitalization (GMD): translation to a novel endoscopic metabolic therapy. Endosc Int Open. 2019 Dec;7(12):E1640-E1645. doi: 10.1055/a-0957-3067. Epub 2019 Nov 25. PMID 31788546
- [Background] Oberbach A, Schlichting N, Kullnick Y, Heinrich M, Lehmann S, Retschlag U, Friedrich M, Fayad L, Dietrich A, Khashab MA, Kalloo AN, Kumbhari V. Gastric mucosal devitalization improves blood pressure, renin and cardiovascular lipid deposition in a rat model of obesity. Endosc Int Open. 2019 Dec;7(12):E1605-E1615. doi: 10.1055/a-0990-9683. Epub 2019 Nov 25. PMID 31788541
- [Background] Itani MI, Oberbach A, Salimian KJ, Enderle M, Hahn H, Abbarh S, Kendrick K, Schlichting N, Anders RA, Besharati S, Farha J, Fayad L, Kalloo AN, Badurdeen D, Kumbhari V. Gastric Mucosal Devitalization (GMD): Using the Porcine Model to Develop a Novel Endoscopic Bariatric Approach. Obes Surg. 2022 Feb;32(2):381-390. doi: 10.1007/s11695-021-05773-4. Epub 2021 Nov 19. PMID 34797503